CLINICAL TRIAL: NCT00183547
Title: Depression Prevention in Pregnant American Indian Teens Using CBT
Brief Title: Depression Prevention Program for American Indian Adolescents During and After Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Golda Ginsburg, PhD, Johns Hopkins Center for American Indian Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R34MH071300 (NIH); R34MH071300 (NIH); DSIR 84-CTP
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2013-05-29 (Estimated); Status verified 2008-12

CONDITIONS: Depression; Pregnancy
Keywords: Postpartum Depression; Postpartum Period; Indians, North American; Adolescent; Female; CBT
MeSH Terms: conditions — Depression; Depression, Postpartum | interventions — Palliative Care

ARMS (2):
- 1 (Experimental): "Living in Harmony" depression prevention program
  Interventions: Behavioral: "Living in Harmony" depression prevention program
- 2 (Active Comparator): Depression-prevention education and support
  Interventions: Behavioral: Depression-prevention education and support

INTERVENTIONS:
Behavioral: "Living in Harmony" depression prevention program — Weekly therapy sessions consisting of cognitive behavioral therapy (CBT), culturally-relevant education, and support
  Arms: 1
Behavioral: Depression-prevention education and support — Weekly therapy sessions offering general depression-prevention education and support
  Arms: 2

SUMMARY:
This study will determine the effectiveness of the "Living in Harmony" depression prevention program in preventing depressive symptoms among pregnant American Indian adolescents during pregnancy and after giving birth.

DETAILED DESCRIPTION:
Pregnancy among reservation-based American Indian adolescents has become increasingly common. Numerous psychosocial and environmental factors have put this population at high risk for pregnancy-related depression. Depression during pregnancy and after giving birth is associated with reduced quality of life for both young mothers and their children. Many reservations lack mental health services; therefore, an inexpensive intervention is needed to prevent depressive symptoms among pregnant adolescents who live on reservations.

The duration of this study will vary for each participant, depending on the time of study entry. Participants will be randomly assigned to receive weekly sessions of either the "Living in Harmony" program, consisting of cognitive behavioral therapy (CBT), culturally-relevant education, and support; or general depression-prevention education and support. Participants' depressive symptoms will be assessed at study entry, at 4, 12, and 24 weeks after giving birth, and study completion. Interviews and self-report scales will be used to assess participants.

ELIGIBILITY:
Inclusion Criteria:

* At 28th week or earlier of pregnancy
* Center for Epidemiologic Studies-Depression Scale (CES-D) score of 16 or higher
* Identified (by others and by self) as an American Indian
* Currently live on an American Indian reservation
* Parent or guardian willing to give consent, if applicable
* Willing and able to comply with all study requirements

Exclusion Criteria:

* Diagnosis of major depressive disorder
* Current psychiatric disorder or condition requiring intervention or treatment
* Current participation in another mental or behavioral health study

Ages: 15 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 45
Dates: Start 2005-01; Primary Completion 2007-03 (Actual); Study Completion 2007-09

PRIMARY OUTCOMES:
Postpartum depression | up to 24 weeks postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Golda Ginsburg, PhD, Principal Investigator — Johns Hopkins Center for American Indian Health
Locations (2):
- United States (2):
  - Johns Hopkins Center for American Indian Health, Whiteriver, Arizona
  - Johns Hopkins Center for American Indian Health, Baltimore, Maryland